## S.A.I.L.I.N.G.

## Studies on Adsorption International Learning Initiative Global

## 1) Research and Researcher's Information

| Research Topic | The use of sorption technologies in patients receiving program hemodialysis with inflammatory syndrome | | | | |
|---|---|---|---|---|---|
| Key Words | Program dialysis Sorption Complications of program dialysis | | Specialty | | Nephrology<br>Blood Purification Therapy |
| Principal<br>Investigator<br>Name | Evgeny Shutov | | Title | | Head of the Nephrology<br>Center, Botkin Hospital, PhD |
| Institute | Botkin Hospital, Moscow | | | | |
| Email | S | nutov_e_v@mail. | ru | Tel. | +79858086519 |
| Address | 125284, M | oscow, 2nd Botki | nsky pr-d, 5 | Code | |
| Research Start and<br>Completion Time | | September 2024<br>August 2025 | | | |

## 2) Research Abstract

| Research Topic | Use of sorption technologies in patients undergoing maintenance hemodialysis with inflammatory syndrome and clinical manifestations of uremia |
|---|---|
| Study Aim | To evaluate the effect of hemosorption with the Jafron HA130 cartridge combined with hemodialysis on inflammatory markers and clinical symptoms of uremic intoxication |
| Study Design | This study will involve 30 hemodialysis patients selected based on examination results showing elevated C-reactive protein (CRP) and/or interleukin-6 (IL-6) levels. Participants will undergo hemoadsorption with the Jafron HA130 cartridge performed concurrently with hemodialysis: three times per week during the first month, twice per week during the second month, and once per week during the third month. The following parameters will be assessed: inflammatory markers (CRP, IL-1, IL-6, IL-8, β2-microglobulin, free light chains of immunoglobulins), parathyroid hormone (PTH), standard biochemical blood tests (creatinine, urea, calcium, phosphorus, albumin, iron metabolism), and complete blood count. Analyses will be performed at baseline (before inclusion) and monthly thereafter. The total study duration will be three months. |
| Total Patient<br>Number | 60 patients |
| | 1. Adequate dialysis defined by a KT/V index ≥ 1.4 |
| | 2. No active inflammatory process or infection |
| Selection of the Patients | 3. Age ≥ 18 years |
| rations | 4. Receiving standard hemodialysis regimen three times weekly, at least 4 hours per session |
| | 5. Elevated interleukin-6 (IL-6) and/or C-reactive protein (CRP) levels above reference values |
| | Exclusive Criteria: |
| | 1. Current use of steroids or immunosuppressive therapy |
| | 2. History of kidney transplantation |
| | Diagnosis of cancer Pregnancy |
| | Intervention Group |

| | Dialysis patients will undergo a combined procedure (hemodialysis and hemosorption) using the Jafron HA130 cartridge three times a week in the first month, twice a week in the next month, once a week in the third month. |
|---|---|
| Treatment Plan | Control Group Patients on standard dialysis procedure (30 patients) |
| Endpoints | Primary Endpoints |
| | The effectiveness of combined procedures (hemodialysis + hemosorption) compared with standard hemodialysis in reducing the level of the IL-6 |
| | Secondary Endpoints |
| | Change from baseline in serum Il-1, IL-8, IL-10, CRP, beta2-microglobulin, free light chains, PTH, serum iron, ferritin, TS, phosphorus, calcium, BUN, creatinine, Hb. |
| | Change from baseline in Hospital Anxiety and Depression Scale Score |
| | Change from baseline in pruritus (Visual Analogue Scale) |
| | Safety Index |
| | Assess safety based on the number of serious adverse events and adverse events |
| Statistics Method | The assessment will be carried out using standard statistical methods |
| Expected Results | Reduced levels of inflammatory markers, middle molecules and associated uremic manifestations |
| The Importance of Study | Improved treatment results |
| Study Duration | 1 year |